CLINICAL TRIAL: NCT03740503
Title: Genomic Investigation of Unusual Responders
Acronym: GENIUS
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: GENIUS
Record Dates: First submitted 2018-10-23; First posted 2018-11-14 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Breast Cancer; Non-small Cell Lung Cancer; Colorectal Cancer; Genitourinary Cancer; Gynecological Cancer; Upper Aerodigestive Tract Cancer; Pancreatobiliary Gastrointestinal Cancer; Melanoma (Skin); Rare Cancer; Carcinoma of Unknown Primary
Keywords: Cancer; Breast Cancer; Non- small Cell Lung Cancer; Colorectal Cancer; Genitourinary Cancer; Gynecological Cancer; Upper Aerodigestive Tract Cancer; Pancreatobiliary Gastrointestinal Cancer; Melanoma Cancer; Rare Cancer; Unknown Primary Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Urogenital Neoplasms; Melanoma; Neoplasms, Unknown Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archival tumor tissue, whole blood at baseline for germ-line DNA analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Studies have shown that tumors from the same patient may respond very differently to the same therapeutic agents. This study aims to investigate the genetic basis of tumors that respond abnormally well or poorly to therapeutic agents in an effort to understand the fundamental genetic basis of this response. The present protocol seeks to retrospectively perform Exome, next-generation (DNA) sequencing and/or other molecular techniques on tumor samples to identify the genetic basis of a patient's exceptional response to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have either an exceptionally good or poor response to treatment, as indicated by their treating physician.

   1. The exact definition of this is adaptable to the disease but a suggested guideline is a Complete Response, Partial Response or progression free interval of at least 6 months
   2. Exceptionally poor response includes patients who were expected to respond favourably to a treatment but instead responded poorly (e.g dramatic tumor growth or death)
2. The patient must have sufficient archival tumor available for sequencing.
3. Deceased patients will also be considered for analysis (up to 30 patients per year) if they meet at least one of the following requirements:

   a)) Patients who have archival tissue stored within the UHN Laboratory Medicine Program who have had a consent waiver granted by the REB to access the tissue.

   b) Patients who have archival tissue banked for further research within the UHN Biospecimen Sciences Program

   Exclusion Criteria:
   * None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled who displayed exceptional response as well as those who were expected to respond favourably but displayed a poor outcome (e.g. drastic tumour growth or death) to their prescribed medication or treatment from a clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-11-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Genomic Characterization of Tumor Samples | Through study completion, up to 2 years
  Characterization of the genetic changes that may explain a tumor's exceptional response or disaster to therapeutc agents.

CONTACTS AND LOCATIONS:
Overall Officials: David Cescon, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Madariaga A, Garg S, Bruce JP, Thiryayi S, Mandilaras V, Rath P, Oza AM, Dhani NC, Cescon DW, Lee YC, Chen E, Wang L, Clarke B, Lheureux S. Biomarkers of outcome to weekly paclitaxel in epithelial ovarian cancer. Gynecol Oncol. 2020 Nov;159(2):539-545. doi: 10.1016/j.ygyno.2020.08.032. Epub 2020 Sep 8. PMID 32912664